CLINICAL TRIAL: NCT03635528
Title: Evaluating Accommodative Responses of Soft Contact Lenses for Myopia Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: CR-6008
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (14):
- Test 1\Test 2\Control 2\Test 3\Control 1\Test 4\Test 5 (Experimental): Subjects between ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 2\Test 3\Test 1\Test 4\Control 2\Test 5\Control 1 (Experimental): Subjects between ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 3\Test 4\Test 2\Test 5\Test 1\Control 1\Control 2 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 4\Test 5\Test 3\Control 1\Test 2\Control 2\Test 1 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 5\Control 1\Test 4\Control 2\Test 3\Test 1\Test 2 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Control 1\Control 2\Test 5\Test 1\Test 4\Test 2\Test 3 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Control 2\Test 1\Control 1\Test 2\Test 5\Test 3\Test 4 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 5\Test 4\Control 1\Test 3\Control 2\Test 2\Test 1 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Control 1\Test 5\Control 2\Test 4\Test 1\Test 3\Test 2 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Control 2\Control 1\Test 1\Test 5\Test 2\Test 4\Test 3 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 1\Control 2\Test 2\Control 1\Test 3\Test 5\Test 4 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 2\Test 1\Test 3\Control 2\Test 4\Control 1\Test 5 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 3\Test 2\Test 4\Test 1\Test 5\Control 2\Control 1 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2
- Test 4\Test 3\Test 5\Test 2\Control 1\Test 1\Control 2 (Experimental): Subjects between the ages of 7 and 25 years will be randomly assigned to one of fourteen unique sequences of the seven lens types.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3; Device: Test Lens 4; Device: Test Lens 5; Device: Control Lens 1; Device: Control Lens 2

INTERVENTIONS:
Device: Test Lens 1 — EMO-114
Device: Test Lens 2 — EMO-116
Device: Test Lens 3 — EMO-118
Device: Test Lens 4 — RMY-100
Device: Test Lens 5 — Biofinity multifocal D Lens
Device: Control Lens 1 — EMO-117
Device: Control Lens 2 — Proclear 1 day

SUMMARY:
This is a bilateral, non-dispensing, randomized, controlled, double-masked, 7x7 cross-over study. Each subject will be bilaterally fitted with one of the 7 test articles in each of the 7 periods for a total of four visits. Up to two lens types will be fit at each of the four study visits.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all following criteria to be enrolled in the study:

  1. Pediatric subjects (<18 years old) must read (or be read to), understand, and sign the Statement of Information and Assent and receive a fully executed copy of the form.
  2. Adult subjects (≥18 years old) and parent(s) or legal guardian(s) of pediatric subjects must read, understand and sign the Statement of Informed Consent and receive a fully executed copy of the form.
  3. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  4. Between 7 and 25 years of age (inclusive).
  5. Have normal eyes (i.e., no ocular medications or infections of any type).
  6. Vertex-corrected distance subjective best-sphere refraction must be between -0.75D and -5.00D (inclusive) in each eye.
  7. Cylindrical refraction must be 1.00D or less in each eye, by subjective sphero-cylindrical refraction.
  8. Have sphero-cylindrical best-corrected visual acuity of 20/25 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any systemic allergies, infectious disease (e.g., hepatitis, tuberculosis, HIV), autoimmune disease (e.g., rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear and/or participation in the study. Specifically, any chronic (3 months or more) or short-term (within 7 days from enrollment) use of oral agents with antimuscarinic properties.
  4. Any current use of ocular topical medication (occasional use of re-wetting drops is allowed). Specifically, any use of topical agents with anti-muscarinic properties within 21 days from enrollment.
  5. Any previous or planned ocular or intraocular surgery, including refractive surgery.
  6. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
  7. Current or recent (within 30 days from enrollment) rigid lens wearers.
  8. History of orthokeratology treatment.
  9. Any known hypersensitivity or allergic reaction to EyeCept® (or sponsor approved equivalent) Rewetting Drop Solution.
  10. Employees or their children/relatives of investigational clinic (e.g., Investigator, Coordinator, Technician).
  11. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to, aphakia, uveitis, ocular hypertension, glaucoma, severe keratoconjunctivitis sicca, history of recurrent corneal erosions, keratoconus, keratoconus suspect, pellucid marginal degeneration, entropion, ectropion, extrusions, chalazia, and recurrent styes.
  12. Any Grade 3 or greater slit lamp findings (eg, edema, corneal neovascularization, corneal staining, tarsal abnormalities, and conjunctival injection) on the FDA scale.
  13. Any ocular abnormality that is contraindicated contact lens wear.
  14. Any corneal scar within central 5mm
  15. Binocular vision abnormality, intermittent strabismus or strabismus.
  16. Any corneal distortion resulting from ocular diseases or previous hard or rigid gas permeable contact lens wear.

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
On-Axis Accommodative Response Method 1 | 10 minutes post-lens insertion
  On-axis accommodative response with target vergence of 0.25D, 1D, 2D, 3D and 4D measured with a wavefront aberrometer.
On-Axis Accommodative Response Method 2 | 10 minutes post lens insertion
  On-axis accommodative response with target vergence of 0.25D, 1D, 2D, 3D and 4D measured with an open-field auto refractor.

SECONDARY OUTCOMES:
Off-Axis Wavefront Aberrations with Accomodation | 10 minutes post-lens insertion
  Off-axis wavefront aberrations at ±10°, ±20°, ±30° retinal eccentricities with targets at 4 meters will be measured.
Off-Axis Wavefront Aberrations without Accomodation | 10 minutes post lens insertion
  Off-axis wavefront aberrations at ±30° retinal eccentricities with targets at 25 cm will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Cheng, Study Chair — Johnson & Johnson Vision Care, Inc.
Locations (1):
- Indiana University, School of Optometry, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No